CLINICAL TRIAL: NCT00662610
Title: A 12-Week, Phase 1, Multicenter, Double-Blind, Randomized, Dose Ranging, Forced Titration, Naproxen-Controlled, Parallel-Group, Pharmacodynamic Study, to Assess the Effects Different Doses of Naproxcinod and Naproxen on Arterial Blood Pressure as Measured by Ambulatory Blood Pressure Monitoring in Osteoarthritis Patients With Controlled Essential Hypertension
Brief Title: A Study to Assess the Effects of Naproxcinod and Naproxen on Blood Pressure Measurements in Osteoarthritis Patients With Controlled High Blood Pressure
Acronym: HCT3012-X-111
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: NicOx, NicOx.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HCT3012-X-111
Record Dates: First submitted 2008-04-16; First posted 2008-04-21 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis; Hypertension
MeSH Terms: conditions — Osteoarthritis; Hypertension | interventions — naproxen-n-butyl nitrate; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- naproxcinod 375 mg - 750 mg -1125 mg bid (Experimental): dose escalating
  Interventions: Drug: naproxcinod 375 mg -750 mg -1125 mg bid
- naproxen 250 mg -500 mg -750 mg bid (Active Comparator): dose escalating
  Interventions: Drug: naproxen 250 mg - 500mg -750 mg bid

INTERVENTIONS:
Drug: naproxcinod 375 mg -750 mg -1125 mg bid — naproxcinod 375 mg -750 mg -1125 mg bid
  Arms: naproxcinod 375 mg - 750 mg -1125 mg bid
Drug: naproxen 250 mg - 500mg -750 mg bid — naproxen 250 mg - 500mg -750 mg bid
  Arms: naproxen 250 mg -500 mg -750 mg bid

SUMMARY:
To assess the effect of naproxcinod vs. naproxen on arterial blood pressure patients with osteoarthritis and controlled essential hypertension

DETAILED DESCRIPTION:
This is a 12-week, randomized, double-blind, multicenter study comparing the effect of naproxcinod and naproxen on 24 hour arterial blood pressure profile. Patients will be randomly allocated to different naproxcinod or naproxen doses in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Men/Women, 40 or older, diagnosed with hip or knee Osteoarthritis.
* Hypertensive patient with treated and controlled essential hypertension.
* Must receive at least one antihypertensive treatment from the following drug classes: Diuretic, Angiotensin-Converting Enzyme (ACE) inhibitor, Angiotensin Receptor Blocker (ARB) or Beta-Blocker (BB).
* Must be current chronic user of NSAIDS or acetaminophen.
* Must discontinue all analgesic therapy at Screening.

Exclusion Criteria:

* More than two different classes of antihypertensive drugs.
* Uncontrolled diabetes.
* Hepatic or renal impairment.
* A history of alcohol/drug abuse.
* Diagnosis of gastric or duodenal ulceration and/or history of significant gastro-duodenal bleeding.
* History of congestive heart failure.
* Clinically relevant abnormal ECG.
* Current or expected use of anticoagulants.
* Current or history of any medical disease that could interfere with the study objectives or put the patient's safety at risk.
* Participation within 30 days prior to pre-screening in another investigational study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To characterize the 24-hour arterial blood pressure profile of different doses of naproxcinod, as measured by ABPM after each treatment period, compared to different doses of naproxen after three 3-week forced titration. | 11 weeks

SECONDARY OUTCOMES:
To evaluate the general safety and tolerability as well as the PK/PD profile of different doses of naproxcinod compared to different doses of naproxen. | 11 weeks

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Mobile, Alabama
  - Tempe, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Buena Park, California
  - Colorado Springs, Colorado
  - Boynton Beach, Florida
  - Stockbridge, Georgia
  - Boise, Idaho
  - Chicago, Illinois
  - Evansville, Indiana
  - Newburgh, Indiana
  - Terre Haute, Indiana
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Billings, Montana
  - Las Vegas, Nevada
  - Edison, New Jersey
  - Binghamton, New York
  - Johnson City, New York
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Clarksville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - Houston, Texas
  - Norfolk, Virginia